CLINICAL TRIAL: NCT05356871
Title: Validity and Reliability of a Clinical Method for Assessment of Cardiorespiratory Fitness Using Seismocardiography
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: VentriJect ApS (Industry)
Responsible Party: Principal Investigator, Jørn Wulff Helge, Professor, University of Copenhagen
Other Study IDs: VentriJect Validation Study
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Cardiorespiratory Fitness Test
Keywords: Validity; Reliability; VO2max testing; Biological age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy participants: Healthy men and women within the age of 18 and 75 yrs.
  Interventions: Other: VO2max validity and reliability assesment

INTERVENTIONS:
Other: VO2max validity and reliability assesment — Reliability assessment of VO2max determination with three repeated measures for two methods.

SUMMARY:
Measurement of cardiorespiratory fitness (here VO2max) is considered a valuable tool for improving the risk prediction of cardiovascular disease and overall patient management. However, the gold standard method for determining VO2max requires both maximal exercise until exhaustion and expensive equipment, why it is not always feasible. A new method for estimating VO2max using a non-exercise prediction model with seismocardiography (SCG) information has been proposed. SCG is recording and interpretations of vibrations originating from the beating heart measured on the chest wall with an accelerometer. SCG has previously been shown to correlate to physiologic events in the cardiac cycle and thus a measure of cardiac performance. VO2max is generally believed to be limited by the rate of oxygen delivery to the muscles, where maximal cardiac output and oxygen carrying capacity of the blood are considered the main limiting factors. The theoretical basis for incorporating SCG to a VO2max prediction model is therefore evident. The previous studies assessed the prediction model in a cross-sectional study design to compare validity of the method. A requirement of further validation of the prediction model with reliability assessment is therefore needed.

Biological age is a concept trying to relate the age to the health status rather than the date of birth. Biological age assesses the heterogeneity in functional metabolic status and vulnerability to disease. A Biological age model has previously been designed for health promotion interventions. However, reliability assessment of the model is needed.

The purpose of the current study was therefore to:

1. investigate the validity and reliability of a new clinical method for estimation of maximal oxygen consumption (VO2max) using seismocardiography.
2. investigate the reliability of the biological age model.

DETAILED DESCRIPTION:
20 healthy participants were recruited for the study. The study included three identical visit to the laboratory within 14 days.

The participants received both written and oral information about the study and the possible risks associated hereof, before volunteering and signing a written informed consent form.

The participants arrived at the laboratory after an overnight fast from latest 10pm the day before (water excepted). Furthermore, the participants were asked to avoid strenuous exercise 48 hours prior to the test day and eat a habitual diet, which had to be replicated before the second and third visit.

Testing at each visit to the laboratory included:

Completion of a short version of the International Physical Activity Questionaire, about leisure time physical activities.

Measurements of height, weight and waist and hip circumference.

Measurement of body composition using a Dual-energy X-ray absorptiometry (DXA) scan on day 1.

Measurement of body composition using a bioelectrical impedance analysis scale on day 1, 2 and 3.

Measurement of blood pressure in the supine position. 3 measures with 2 minute resting in between.

Measurement of VO2max using a non-exercise testing method based on seismocardiography.

Collection of a 15 ml resting venous blood sample for measurements of resting levels of hormones, metabolites and lipids in the blood plasma.

Measurement of lung function in terms of FEV1 and FVC (Vyntus SPIRO spirometer, Vyaire Medical).

Determination of VO2max applying a graded exercise test on a bicycle ergometry until voluntary exhaustion with continuous pulmonary gas exchange measurements.

Procedure and analysis:

Bioelectrical impedance analysis scale (Tanita MC-780MA, Tanita Corporation of America Inc): The participants was analysed on the scale after voiding and wearing minimal clothing.

DXA scanning (Lunar iDXA, GE Healthcare): The participants was placed in the supine position in the DXA scanner after voiding and while wearing minimal clothing.

Blood samples: The blood samples was collected from the vein cubiti medialis in the forearm. The blood was sampled in iced BD vacutainers (5 mL Aprotinin, 4 mL EDTA and 2 mL Lithium Heparin) and immediately centrifuged at 4000 g for 10 minutes at 4⁰C (Rotina 380R, Hettich). The plasma was collected and stored at -80⁰C for later analyzes of resting levels of metabolites, lipids and hormones.

The concentrations of hemoglobin, hematocrit, glucose and lactate was immediately analyzed though sampling of 2 mL blood in a specialized syringe (safePICO Aspirator, Radiometer) and using an automatic analyzer (ABL800 Flex, Radiometer).

SCG VO2max prediction:

The SCG VO2max prediction was performed as previously described with the same type of equipment. Brief, the SCG recording was performed using an iWorx IX-228/s (IWORX, Dover, New Hampshire) connected to a PC. LabScribe was used as recording software (version 3. Dover, New Hampshire). The accelerometer (Silicon Design 1521-002) had a resolution of ± 2 g, a low noise at 7 μg / √ Hz and a frequency 70 response of 0-300 Hz and was placed on sternum 2 cm proximal of processus xiphoideus. The recording lasted 5 minutes and was performed in the supine position. VentriJect Aps later performed the signal processing and VO2max estimation. VentriJect Aps was informed of the age, height and weight of the participants for inclusion in the prediction model, but was blinded of the measured VO2max.

Hereafter a new devolved wireless device (Seismofit, VentriJect Aps) was used to determine SCG VO2max. The Seismofit contains a 3v battery and a three-axis digital output accelerometer (LIS3DHH, ST Microelectronics). The Seismofit device is connected to a phone application where the participants demographic data (age, height and weight) was entered before performing the recording. For the recording, the participants was lying in the supine position and the Seismofit device was placed on sternum 2 cm proximal of processus Xiphoideus with double adhesive tape. The predicted SCG VO2max value appeared on the phone screen within 5 minutes.

The Seismofit VO2max prediction was performed twice with 5 minutes rest in between. This was done to assess the test-retest reliability of the device.

The iWorx VO2max was done to compare the previous equipment with the new wireless equipment with automatic signal processing.

The gold standard VO2max determination:

A graded exercise test (GET) until voluntary exhaustion on a bicycle ergometer was performed. The protocol consisted of a five-minute warm-up at 80 W for women and 100 W for men and increased hereafter with 20 W for women and 25 W for men every minute until exhaustion.

Participants was wearing a chest strapped heart rate monitor (Polar Vantage XL, Polar) with continuous heart rate measures during the test. Furthermore the participants, was asked about perceived exhaustion on the 6-20 Borg scale directly following exhaustion.

Statistical analysis:

All data was checked for normal distribution (Shapiro-Wilk test) and equal variance (Brown- Forsythe test). The significant level is p<0.05.

A Mixed-effect model, Bland-Altman analysis with 95% limits of agreement, Pearson correlations and Mean Absolute Percentage Error was used for assessment of validity between the Seismofit VO2max and GET VO2max, Seismofit VO2max measure 1 and 2 and between Seismofit VO2max and iWorx VO2max.

Coefficient of Variation (CV), Standard Error of Estimate (SEE) and Intraclass Correlation Coefficient (ICC) was used to assess reliability of VO2max measurements.

The project was approved by the Science Ethical commitee of the greater region of Copenhagen (H-19081375) the 3rd of February 2020. The protocol of the study adhered to the principles of the Helsinki declaration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants

Exclusion Criteria:

* A history of previous or current cardiovascular disease
* Pregnancy
* Conditions that prevent maximal cycling exercise

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A representative selection of the healthy adult population
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Validity and reliability of the SCG VO2max prediction model | From June until December
  For assessment of validity and reliability of the SCG VO2max prediction model, three repeated measures of SCG VO2max and the gold standard determination of VO2max will be conducted on three different test days within 14 days.
  The validity assessment will be based on differences and agreement between the two methods.
  The reliability assessment will be based on intra-method variations between test days.

SECONDARY OUTCOMES:
Reliability of the biological age model | From June until December
  Three repeated measures of biological age within 14 days will be conducted.
  The reliability assessment will be based on intra-method variation between test days

CONTACTS AND LOCATIONS:
Overall Officials: Jørn W Helge, Professor, Principal Investigator — Department of Biomedical Sciences, Faculty of Health and Medical Sciences, University of Copenhagen
Locations (1):
- Xlab, Faculty of Health and Medical Sciences, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sorensen K, Schmidt SE, Jensen AS, Sogaard P, Struijk JJ. Definition of Fiducial Points in the Normal Seismocardiogram. Sci Rep. 2018 Oct 18;8(1):15455. doi: 10.1038/s41598-018-33675-6. PMID 30337579
- [Background] Sorensen K, Poulsen MK, Karbing DS, Sogaard P, Struijk JJ, Schmidt SE. A Clinical Method for Estimation of VO2max Using Seismocardiography. Int J Sports Med. 2020 Sep;41(10):661-668. doi: 10.1055/a-1144-3369. Epub 2020 May 26. PMID 32455456
- [Background] Hansen MT, Grønfeldt BM, Rømer T, Fogelstrøm M, Sørensen K, Schmidt SE, et al. Determination of Maximal Oxygen Uptake Using Seismocardiography at Rest. In: Computing in Cardiology 2021. IEEE. 2021;48(1):48-51 DOI: 10.22489/CinC.2021.165
- [Background] Husted KLS, Fogelstrom M, Hulst P, Brink-Kjaer A, Henneberg KA, Sorensen HBD, Dela F, Helge JW. A Biological Age Model Designed for Health Promotion Interventions: Protocol for an Interdisciplinary Study for Model Development. JMIR Res Protoc. 2020 Oct 26;9(10):e19209. doi: 10.2196/19209. PMID 33104001